CLINICAL TRIAL: NCT01844973
Title: Study to Evaluate the Pharmacokinetics and the Safety of M518101 in Plaque Psoriasis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho North America Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: M518101-US05
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle
- M518101 (Active Comparator)
  Interventions: Drug: M518101

INTERVENTIONS:
Drug: M518101 — Proper quantity twice a day
  Arms: M518101
Drug: Vehicle — Proper quantity twice a day
  Arms: Vehicle

SUMMARY:
This study is to evaluate the pharmacokinetics and safety of M518101 in male and female plaque psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

* Who are able and willing to give signed informed consent
* Who are male or females aged 18 years or older with plaque psoriasis confirmed by the Investigator.
* Who have ≥20% of body surface area (BSA) afflicted with plaques
* Who are neither pregnant nor breast-feeding, nor plan to become pregnant during the study.

Exclusion Criteria:

* Who have a history of allergy to vitamin D3 derivative preparations or a history of relevant drug hypersensitivity.
* BMI > 32.0 kg/m2
* Who are pregnant or lactating.
* Who have any renal or hepatic insufficiency, or clinically significant cardiac, renal or hepatic disease.
* Who are not deemed eligible as determined by medical history, physical examination or clinical laboratory safety tests.
* Who have clinically relevant history or presence of any disease or surgical history other than psoriasis which is likely to affect the conduct of the study.
* Whose serum calcium levels exceed the upper limit of reference range
* Who have used any investigational medicinal product and/or participated in any clinical study within 60 days of randomization.
* Who have taken any durg with known effects on calcium metabolism within 30days of randomization
* Who have been treated with any drug with a known risk of QT prolongation within 30days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of M5181 | 0, 1, 2, 4, 6, 9 12h after dosing
Peak Plasma concentration (Cmax) of M5181 | 0, 1, 2, 4, 6, 9 12h after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Orenge County Research Center, Tustin, California, United States